CLINICAL TRIAL: NCT02530632
Title: The Effects of General Anesthesia on Microcirculation of Central and Peripheral Soft Tissue: a Comparison of Inhalational and Intravenous Anesthetics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 201504089RIND
Record Dates: First submitted 2015-08-17; First posted 2015-08-21 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Microcirculatory Effects of Anesthesia; Inhalation and Intravenous Anesthesia
Keywords: microperfusion; temperature; near-infrared spectroscopy; anesthesia; total intravenous anaesthesia
MeSH Terms: conditions — Respiratory Aspiration | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane anesthesia (Active Comparator): Anesthesia maintained with inhalational sevoflurane
  Interventions: Drug: Sevoflurane; Procedure: General anesthesia induction
- Propofol anesthesia (Experimental): Anesthesia maintained with intravenous propofol continuous infusion
  Interventions: Drug: Propofol; Procedure: General anesthesia induction

INTERVENTIONS:
Drug: Propofol — General anesthesia maintained with intravenous propofol infusion
  Arms: Propofol anesthesia
Drug: Sevoflurane — General anesthesia maintained with inhalational sevoflurane
  Arms: Sevoflurane anesthesia
Procedure: General anesthesia induction — Induce routine of general anesthesia, including propofol 1-3mg/kg, fentanyl 1-3mcg/kg, cisatracurium 0.2-0.3mg/kg.

SUMMARY:
Effects of different general anesthetics on peripheral microcirculation.

DETAILED DESCRIPTION:
Human keep body temperature in a narrow range by a variety of regulatory mechanism. Peripheral thermal receptors send signals to central nervous system which regulate body temperature via peripheral effectors, such as vasoconstriction, vasodilatation, shivering, sweating and etc. In patients undergoing general anesthesia, the regulatory mechanism is altered. General anesthesia changes blood distribution in the body, the metabolic rate of muscle, threshold of thermal regulation in the brain and etc, so that heat distribution and microcirculation condition will also change. In this study, near-infrared spectroscopy (NIRS) is used to measure the microcirculatory condition. NIRS is a non-invasive continuous measurement to detect tissue saturation with the method of different wavelength of near-infrared. General anesthesia with inhalational sevoflurane and intravenous propofol is separated into 2 groups. Because of different mechanism of general anesthesia of these 2 anesthetics, different physiologic response may occur. Body temperature and somatic saturation are compared in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Breast surgeries under general anesthesia
2. BMI 18.5~30

Exclusion Criteria:

1. Cardiac disease
2. Lung disease
3. Renal disease
4. Neurological disease
5. Autonomic nervous system dysfunction

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Somatic saturation | during surgery, approximately 2-4 hr
  Change of somatic saturation measured by NIRS

SECONDARY OUTCOMES:
Body temperature | during surgery, approximately 2-4 hr
  Nasal and peripheral temperature

CONTACTS AND LOCATIONS:
Overall Officials: Shou-Zen Fan, Principal Investigator — Department of Anesthesiology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan